CLINICAL TRIAL: NCT00012675
Title: Developing and Implementing a Quality Measure for Glycemic Control
Status: Withdrawn | Type: Observational
Why Stopped: This study was withdrawn prior to enrollment.
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: DII 99-205
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2012-05-24 (Estimated); Status verified 2012-05

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1

SUMMARY:
Many patients with diabetes are under sub-optimal glycemic control. Central to the clinician's task in improving glycemic control is the management of hypoglycemic medication therapy, including the use of drugs such as insulin and sulfonylureas. Clinical trials have demonstrated that more intensive hypoglycemic medication therapy results in improved glycemic control. Yet quality measures for this critical process of care have not been developed and we know little about how physicians actually manage hypoglycemic medications.

DETAILED DESCRIPTION:
Background:

Many patients with diabetes are under sub-optimal glycemic control. Central to the clinician's task in improving glycemic control is the management of hypoglycemic medication therapy, including the use of drugs such as insulin and sulfonylureas. Clinical trials have demonstrated that more intensive hypoglycemic medication therapy results in improved glycemic control. Yet quality measures for this critical process of care have not been developed and we know little about how physicians actually manage hypoglycemic medications.

Objectives:

We propose to develop a quality measure that describes the intensity of physicians' hypoglycemic medication therapy. We will then provide feedback to VA physicians regarding their practices and access to experts in diabetes care to determine whether this intervention leads to improvements in glycemic control.

Methods:

The study was divided into two phases. During the first phase we used existing data to model the decision to increase hypoglycemic medications. At each medical visit, we determined whether an increase in medication therapy occurred. We then used recursive partitioning to develop a model that identified patient characteristics at the visit, such as recent laboratory results and diagnoses, associated with the decision to increase therapy. This model assigns a predicted probability of an increase in therapy to each visit. We used these predictions to define an intensity of hypoglycemic medication therapy for each physician that compared the actual to predicted number of increases over all patient-visits. The second phase was a randomized trial in which clinicians at experimental sites receive feedback on performance and access to expert opinion while usual care is provided at control sites. Feedback on performance was provided twice over 6 months. The change in intensity of treatment scores and glycosylated hemoglobin levels pre- and post-intervention at these sites were compared to performance of primary care physicians at control sites not receiving the intervention.

Status:

Completed.

ELIGIBILITY:
Inclusion Criteria:

Clinic patients with diabetes

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Study Completion 2003-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan R. Berlowitz, MD MPH, Principal Investigator — Bedford VA Medical Center
Locations (1):
- Bedford VA Medical Center, Bedford, Massachusetts, United States

REFERENCES:
- [Result] Berlowitz DR, Ash AS, Glickman M, Friedman RH, Pogach LM, Nelson AL, Wong AT. Developing a quality measure for clinical inertia in diabetes care. Health Serv Res. 2005 Dec;40(6 Pt 1):1836-53. doi: 10.1111/j.1475-6773.2005.00436.x. PMID 16336551
- [Result] Chaudhry SI, Berlowitz DR, Concato J. Do age and comorbidity affect intensity of pharmacological therapy for poorly controlled diabetes mellitus? J Am Geriatr Soc. 2005 Jul;53(7):1214-6. doi: 10.1111/j.1532-5415.2005.53370.x. PMID 16108941
- [Result] Pugh MJ, Anderson J, Pogach LM, Berlowitz DR. Differential adoption of pharmacotherapy recommendations for type 2 diabetes by generalists and specialists. Med Care Res Rev. 2003 Jun;60(2):178-200. doi: 10.1177/1077558703060002003. PMID 12800683